CLINICAL TRIAL: NCT00929929
Title: Randomized Double-blind, Placebo-controlled, Parallel Design, Pilot Study to Assess the Effect of a Nutritional Supplement With Leucine, Along With a Progressive Resistance Exercise Program, on Muscle Strength and Quality of Life in Elderly People.
Brief Title: Study to Assess the Effect of Leucine Along With Resistance Exercise on Muscle Strength and Quality of Life in Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Pere Leyes, Specialist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRA_LEU-09
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Ageing
Keywords: Aging; Functionality; Sarcopenia; Leucine; Progressive resistance exercise
MeSH Terms: conditions — Sarcopenia | interventions — Leucine; maltodextrin; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Leucine (Experimental): This arm receives a supplement of leucine along with a progressive resistance exercise program.
  Interventions: Dietary Supplement: L-leucine.; Behavioral: Exercise program.
- Maltodextrin (Placebo Comparator): This arm receives a supplement of maltodextrin along with a progressive resistance exercise program.
  Interventions: Dietary Supplement: Maltodextrin.; Behavioral: Exercise program.

INTERVENTIONS:
Dietary Supplement: L-leucine. — 10 g of leucine per day, during 12 weeks.
  Other Names: Leucine.
  Arms: L-Leucine
Dietary Supplement: Maltodextrin. — 10 g of maltodextrin per day, during 12 weeks.
  Other Names: Maxijul.
  Arms: Maltodextrin
Behavioral: Exercise program. — Progressive resistance exercise program 4 days a week, during 12 weeks.
  Other Names: Resistance exercise.

SUMMARY:
The purpose of this study is to determine whether a nutritional supplement with an amino acid called leucine along with resistance exercise are effective in the improvement of muscle strength and quality of life in elderly people.

DETAILED DESCRIPTION:
Physiological aging is accompanied by functional loss and changes in different organs, including the skeletal muscle, with a progressive reduction in muscle mass. This is called physiological sarcopenia of the elderly.

In any population of autonomous individuals over 65 years, a proportion between 3% and 32% depending on age, meets the criteria of the so-called Frailty Syndrome. Frailty is characterized by a decrease in reserves and resistance to aggression, conferring increased vulnerability, disability and poor vital prognosis.

A feature of the Frailty Syndrome is the potential reversibility of many of the elements at the initial stages of frailty. Currently, available treatment for frailty is limited. One of the tools should be the prevention of sarcopenia, where nutritional treatment and exercise have a vital role.

Protein synthesis in aged muscle can be improved by increasing leucine concentration above physiological levels by a higher intake. Regarding exercise, progressive resistance training is one of the interventions that have shown better results in the increase of mass and muscle strength in elderly people.

The hypothesis raises the possibility that an intervention consisting of a leucine supplement along with progressive resistance training, is superior to the same training program and a placebo in improving muscle strength and quality of life in elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Over 70 years of age.
* Subjects capable of doing resistance exercise.

Exclusion Criteria:

* Hospitalized patients.
* Disabled patients (i.e., not being able to exercise).
* Patients that usually train in resistance exercise.
* Patients with chronic renal failure.
* Patients with a fractured extremity during the last 6 months.
* Patients that follow diets with a protein restriction.
* Patients with oral nutritional support, enteral or parenteral nutrition.
* Patients in a low calorie diet to lose weight.
* Patients using pharmacological treatment with anorexigenic effects, anabolic steroids or corticosteroids.
* Patients with cognitive impairment or major psychiatric disorder.
* Non-signed informed consent.
* Any patient not capable to properly follow the treatment or not considered adequate by the researchers.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Muscle strength. | Baseline, 4 weeks, 12 weeks

SECONDARY OUTCOMES:
Functionality | Baseline, 4 weeks, 12 weeks

OTHER OUTCOMES:
Quality of life | Baseline, 4 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Forga, MD, Principal Investigator — Hospital Clinic of Barcelona; Joan Trabal, RD, MS, Study Chair — Hospital Clinic of Barcelona; Pere Leyes, MD, Study Chair — Hospital Clinic of Barcelona; Andreu Farran, PhD, Study Chair — University of Barcelona
Locations (1):
- Nutrition and Dietetics Unit, Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- See also: A brief definition of the Frailty Syndrome. — http://en.wikipedia.org/wiki/Frailty_syndrome